CLINICAL TRIAL: NCT01387698
Title: Observatoire Prospectif, Longitudinal Dans la Prise en Charge Thérapeutique de La Rectocolite Hémorragique légère à Modérée
Brief Title: Prospective, Longitudinal Multicentric Survey in the Therapeutic Care of Mild to Moderate Ulcerative Colitis
Acronym: OPTIMUM
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: FE999907 CS09
Record Dates: First submitted 2011-06-29; First posted 2011-07-04 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study is to confirm the long-term efficacy (remission and maintenance in remission) of current validated treatments. Each patient will be followed during 3 years in this non-interventional trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or above
* Ulcerative colitis, whatever the extension, in mild to moderate flare-up (including proctitis)
* Having received the information sheet

Exclusion Criteria:

* Participating, at the time of inclusion, in another study using an investigational drug or device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients at least 18 years old suffering from mild to moderate active ulcerative colitis (whatever the extension)
Sampling Method: Non-Probability Sample
Enrollment: 812 (Actual)
Dates: Start 2011-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Remission rate (ulcerative colitis) - calculated by UCCS (Ulcerative Colitis Clinical Score) | From baseline (inclusion visit) and at 1 year interval after baseline
Remission rate (ulcerative colitis) - calculated by UCCS (Ulcerative Colitis Clinical Score) | From baseline (inclusion visit) and at 2 year interval after baseline
Remission rate (ulcerative colitis) - calculated by UCCS (Ulcerative Colitis Clinical Score) | From baseline (inclusion visit) and at 3 year interval after baseline

SECONDARY OUTCOMES:
Remission rate (endoscopic) - calculated by UC-DAI (Ulcerative Colitis Disease Activity Index) | From baseline (inclusion visit) and at 1 year interval after baseline
Assessing treatment adherence by patient's completion of questionnaire MMAS-8 (Modified Morisky Adherence Scale) | From baseline (inclusion visit) and at 1 year interval after baseline
Occurence/number of adverse events | From baseline (inclusion visit) to year 3 after baseline
Colonoscopy (if available) - assessing endoscopic activity of the ulcerative colitis | From baseline (inclusion visit) to 3 year after baseline
Remission rate (endoscopic) - calculated by UC-DAI (Ulcerative Colitis Disease Activity Index) | From baseline (inclusion visit) and at 2 year interval after baseline
Remission rate (endoscopic) - calculated by UC-DAI (Ulcerative Colitis Disease Activity Index) | From baseline (inclusion visit) and at 3 year interval after baseline
Assessing treatment adherence by patient's completion of questionnaire MMAS-8 (Modified Morisky Adherence Scale) | From baseline (inclusion visit) and at 2 year interval after baseline
Assessing treatment adherence by patient's completion of questionnaire MMAS-8 (Modified Morisky Adherence Scale) | From baseline (inclusion visit) and at 3 year interval after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (158):
- France (158):
  - Centre Hospitalier pays d aix, Aix-en-Provence
  - Investigational site, Amboise
  - Cabinet Médical, Amiens
  - CMAD, Amiens
  - Clinique Saint Joseph, Angers
  - Investigational site, Anglet
  - Cabinet Médical, Arras
  - Hopital Robert Ballanger, Aulnay-sous-Bois
  - Investigational site, Aulnays Sous Bois
  - Polyclinique Ste Marguerite, Auxerre
  - Investigational site, Beausoleil
  - Clinique ANNE D'ERTOIS, Béthune
  - Le Rabelais, Béziers
  - Centre Hospitalier de Blois, Blois
  - Investigational site, Bordeaux
  - CH de Bourg-en Bresse Hopital de Fleyriart (Viriat), Bourg-en-Bresse
  - Polyclinique Jean Villar, Bruges
  - Cabinet Médical, Caen
  - Cabinet Medical, Cahors
  - Polyclinic Montréal, Carcassonne
  - Investigational site, Carpentras
  - Maison de Consultations, Cesson-Sévigné
  - Investigational site, Challes-les-Eaux
  - CH de Chambery, Chambéry
  - Pole Santé Léonard de Vinci, Chambray-lès-Tours
  - Cabinet Médical, Charleville-Mézières
  - Centre Hospitalier du Haut Anjou Hospital St Julien, Château-Gontier
  - Cabinet Médical, Châteaubriant
  - Cabinet Médical, Châteauroux
  - CH Chateauroux, Châteauroux
  - Hospital, Châteauroux
  - Investigational site, Châteauroux
  - Cabinet Médical, Cherbourg
  - Investigational site, Chinon
  - Cabinet Médical, Clermont-Ferrand
  - Cabinet Médical, Colombes
  - Clinique des Cèdres, Cornebarrieu
  - Centre Hospitalier LAENNEC, Creil
  - CHI Créteil, Créteil
  - Hospital, Créteil
  - Investigational site, Créteil
  - Cabinet Médical, Dax
  - Cabinet Médical, Décines-Charpieu
  - Investigational site, Dijon
  - Investigational site, Dole
  - Octogone, Draguignan
  - Hospital De Dreux, Dreux
  - Hopital Simone Veil, Eaubonne
  - Cabinet Médical, Échirolles
  - Clinic De La Présentation, Fleury-les-Aubrais
  - Centre Hospitalier du Val d'Ariège, Foix
  - Investigational site, Fontenay-le-Comte
  - Investigational site, Gien
  - Cabinet Médical, Grenoble
  - Investigational site, Guigamp Pabu
  - Investigational site, Irigny
  - Cabinet Médical, La Chaussée-Saint-Victor
  - Sarthe et Loir / Médecine IV Hospital, La Flèche
  - Centre Hospitalier Departemental Les Oudairies, La Roche-sur-Yon
  - Hospital Les Oudairies, La Roche-sur-Yon
  - Cabinet Médical, La Varenne-Saint-Hilaire
  - CH Lagny Marne La Vallee, Lagny-sur-Marne
  - Clinique St Ame, Lambres-lez-Douai
  - Investigational site, Lannion
  - Investigational site, Le Cannet
  - Clinique bon Secours, Le Puy-en-Velay
  - Cabinet Médical, Lille
  - Investigational site, Limoges
  - Polyclinique de Lisieux, Lisieux
  - Investigational site, Lorient
  - Hopital Prive Jean Mermoz, Lyon
  - Hopital Privé Jean Mermoz, Lyon
  - Cabinet Médical, Marseille
  - Hopital Clinique Claude Bernard, Metz
  - HPM Site Sainte-Andre, Metz
  - Private hospital of Metz, Metz
  - CHG Montauban, Montauban
  - Centre Hospitalier Montelimard, Montelimard Cedex
  - Cabinet Médical, Montelimard
  - Centre Hospitalier Montélimard, Montelimard
  - Investigational site, Montelimard
  - CHI Le Raincy Montfermeil, Montfermeil
  - Hospital Le Raincy Montfermeil, Montfermeil
  - Cabinet Médical, Montpellier
  - Hopital Saint Eloi, Montpellier
  - Hospital Saint Eloi, Montpellier
  - Investigational site, Montrouge
  - Cabinet Médical, Mulhouse
  - Centre Erdre-Saint Augustin, Nantes
  - Centre Medical Erdre-St Augustin, Nantes
  - Centre Médical Erdre-St Augustin, Nantes
  - Investigational site, Narbonne
  - Cabinet Médical, Nice
  - CHU de Nice-Hopital de l'Archet, Nice
  - Investigational site, Nice
  - Investigational site, Niort
  - Cabinet Médical, Nîmes
  - Le Méridien, Nîmes
  - Hopital de Guingamp, Pabu
  - Cabinet Médical, Paris
  - Clinique du Louvre, Paris
  - Investigational site, Paris
  - Centre Hospitalier de Perpignan, Perpignan
  - Cabinet Médical, Prades
  - Centre Hospitalier d'Annecy, Pringy
  - Cabinet Médicale, Quévert
  - Investigational site, Reims
  - Clinique La Sagesse, Rennes
  - Investigational site, Riom
  - Investigational site, Rodez
  - Clinique de l'Europe, Rouen
  - Clinique Mathilde, Rouen
  - Investigational site, Saint-Brieuc
  - Centre Hospitalier Prive Saint Gregoire, Saint-Grégoire
  - Centre Hospitalier Privé Saint Gregoire, Saint-Grégoire
  - Centre Médical des Châtaigniers, Saint-Herblain
  - Investigational site, Saint-Jean-de-Luz
  - Cabinet Médical, Saint-Jean-de-Védas
  - Investigational site, Saint-Lô
  - Cabinet Lamartine, Saint-Nazaire
  - Polyclinique de l'Ocean, Saint-Nazaire
  - Polyclinique de l'Océan, Saint-Nazaire
  - Investigational site, Saint-Quentin
  - Investigational site, Saint-Raphaël
  - Cabinet Médical, Sarreguemines
  - Investigational site, Sarreguemines
  - Cabinet Médical, Saumur
  - Cabinet Médical, Savigny-sur-Orge
  - Cabinet Médical, Sevran
  - Cabinet Médical, Strasbourg
  - Cabinet Médical, Sucy-en-Brie
  - Investigational site, Tarbes
  - Investigational site, Thionville
  - Cabinet Médical, Toulon
  - Clinic Saint Jean Languedoc, Toulouse
  - Investigational site, Toulouse
  - Cabinet Médical, Tourcoing
  - Centre Hospitalier de Tourcoing-Hôpital DRON, Tourcoing
  - Investigational site, Tournefeuille
  - Cabinet Médical, Troyes
  - Centre Hospitalier de Valence, Valence
  - Clinic, Valence
  - Hospital of Valence, Valence
  - Centre Hospitalier de Valenciennes, Valenciennes
  - Investigational site, Vannes
  - Cabinet Médical, Vendôme
  - Centre Futura Medica, Verguigneul
  - Investigational site, Vernon
  - Cabinet Médical, Vesoul
  - Groupe hospitalier les Portes du Sud, Vénissieux
  - Groupe Hospitalier Mutualiste "Les Portes du Sud", Vénissieux
  - Groupe Hospitalier Mutualiste Les Portes du Sud, Vénissieux
  - Centre Chirurgical St laurent, Villemoisson-sur-Orge
  - CH Villeneuve Saint Georges, Villeneuve-Saint-Georges
  - CHIV, Villeneuve-Saint-Georges
  - Hospital of Villeneuve Saint Georges, Villeneuve-Saint-Georges
  - Cabinet Médical, Vincennes
  - Investigational site, Vincennes